CLINICAL TRIAL: NCT05284227
Title: Artificial Intelligence-augmented Perioperative Clinical Decision Support
Acronym: KIPeriOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Goethe University (Other); Charite University, Berlin, Germany (Other); Asklepios Kliniken Hamburg GmbH (Other); Fraunhofer Institute for Digital Medicine MEVIS (Unknown); Technical University of Munich (Other); RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KIPeriOP 2022
Record Dates: First submitted 2022-02-21; First posted 2022-03-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: ASA Class III/IV Patients; Surgery; Clinical Decision Support Systems
Keywords: Anaesthesiology; Clinical Decision Support; Artificial Intelligence; Perioperative Risk Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Decision Support Application guided Anaesthesiological Assessment (Active Comparator): Preoperative anaesthesiological assessment and risk evaluation using a clinical decision support application.
  Interventions: Other: Electronic Clinical Decision Support Application
- Standard Anaesthesiological Assessment (Sham Comparator): Preoperative anaesthesiological assessment using standard procedures of the hospital and a sham clinical decision support application.
  Interventions: Other: Standard procedures of the hospital and Sham Clinical Decision Support Application

INTERVENTIONS:
Other: Electronic Clinical Decision Support Application — Preoperative anaesthesiological assessment and risk evaluation using a clinical decision support application, that calculates perioperative risks for the patient and informs the anaesthesiologist on indicated diagnostics and procedures according to clinical guidelines in real-time.
  Arms: Clinical Decision Support Application guided Anaesthesiological Assessment
Other: Standard procedures of the hospital and Sham Clinical Decision Support Application — Preoperative anaesthesiological assessment using standard procedures of the hospital. In addition a sham clinical decision support application will be used. Information on perioperative risks and indicated diagnostic procedures according to clinical guidelines is not given to the physician.
  Arms: Standard Anaesthesiological Assessment

SUMMARY:
The study investigates a novel anaesthesiological clinical decision support (CDS) application, that integrates risk evaluation tools and updated clinical guidelines guided by artificial intelligence in the setting of preoperative anaesthesiological assessment. It will be compared to the current standard preoperative assessment workflow with participants being actual patients. 480 participants will be randomly assigned to either the CDS group (preoperative assessment using the CDS application) or the Control group (standard preoperative assessment workflow).

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anaesthesiologists)-Class III and IV
* non-cardiac surgery

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Number of clinically not indicated preoperative diagnostic procedures ordered by the anaesthesiologist | preoperative assessment until operative procedure
  Preoperative diagnostic procedures ordered by the anaesthesiologist are defined as ECG, echocardiography, carotid (Duplex) ultrasound, chest X-ray and functional non-invasive tests for coronary artery disease (e.g. stress echocardiography)

SECONDARY OUTCOMES:
Number of documented items from a predefined set of relevant cardiovascular symptoms and conditions during the anaesthesiological assessment | preoperative assessment until operative procedure
  Completeness of medical documentation will be measured by the number of documented items from a predefined list of relevant cardiovascular symptoms and conditions during the preoperative anaesthesiological asssessment.
Incidence of intra- and postoperative complications | operative procedure until hospital discharge, assessed up to 4 weeks
Incidence of 30-Day unplanned All-cause Hospital Readmission | hospital discharge until 30th postoperative day
Length of Hospital Stay | hospital admission until hospital discharge, assessed up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, M.D., Principal Investigator — Wuerzburg University Hospital
Locations (1):
- University Hospital Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No